CLINICAL TRIAL: NCT07007013
Title: Impact of Humor Prescription on the Emotional Well-being of Patients With Medically Unexplained Symptoms: A Quasi-experimental Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSAPG-75
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Medically Unexplained Symptoms
Keywords: Medically unexplained symptoms
MeSH Terms: conditions — Medically Unexplained Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- humor therapy (Experimental): All participants will receive an intervention based on humor therapy
  Interventions: Other: Humor therapy

INTERVENTIONS:
Other: Humor therapy — The intervention consists of a cycle of 8 group sessions (one per week) led by trained professionals specialized in humor ('clown doctors'). Each session will last approximately 90 to 120 minutes

SUMMARY:
This study aims to study the effectiveness of the intervention for medically unexplained symptoms(MUS) in terms of changes in emotional well-being before and after the intervention (humor therapy)

ELIGIBILITY:
Inclusion Criteria:

* Participants may be included in the trial if they meet all of the following inclusion criteria:
* Men and women over 18 years of age.
* Diagnosed with the condition under study (see Section 2: Definitions).
* Expected to undergo follow-up for their condition at the study center.
* Ability to participate in the required assessments.
* Legal capacity to provide informed consent.
* Signed informed consent for inclusion in the study, either by the participant or their legal representative.

Exclusion Criteria:

* Participants will be excluded if they meet any of the following exclusion criteria:
* Participants diagnosed with any of the following conditions:
* Severe mental health disorder, as determined by the investigator
* Cognitive impairment of any etiology, as recorded in the medical history
* Treatment for the condition under study using community-based resources prescribed in Primary Care within the past 6 months.
* Cognitive or affective disorders that limit the ability to comply with study procedures.
* Participation in another study involving an experimental intervention during the period of the present trial and/or requiring visit schedules that are incompatible with this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
emotional well-being | From baseline to 6 months after ending the intervention
  Emotional well-being will be measured before-after intervention through the Warwick-Edinburgh Mental Well-being Scale (WEMWBS). Range scale: 14-70. Higher scores indicate greater well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Sarai Cuevas, Principal Investigator — CSAPG
Locations (1):
- CAPI Baix A Mar (CSAPG), Vilanova i la Geltrú, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.